CLINICAL TRIAL: NCT02701127
Title: Molecular Effects of Vitamin B3 (Niacinamide) in Acute Kidney Injury
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Ali Poyan Mehr, Instructor in Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2016P000028
Record Dates: First submitted 2016-02-29; First posted 2016-03-08 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Niacinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Niacinamide 1 gram (Active Comparator): Oral niacinamide, 1 gram daily
  Interventions: Drug: Oral niacinamide, 1 gram daily
- Niacinamide 3 grams (Active Comparator): Oral niacinamide, 3 grams daily
  Interventions: Drug: Oral niacinamide, 3 gram daily
- Placebo (Placebo Comparator): Oral placebo pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral niacinamide, 1 gram daily
  Arms: Niacinamide 1 gram
Drug: Oral niacinamide, 3 gram daily
  Arms: Niacinamide 3 grams
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a single center, randomized, single-blind, placebo-controlled study to evaluate the safety and biochemical effects of niacinamide on metabolic parameters of the kidney in patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion criteria

1. All patients undergoing cardiac surgery with the use of cardiopulmonary bypass at high risk for acute kidney injury. A Cleveland score of 6 or more is used to define patients at high risk for acute kidney injury
2. Age ≥ 18
3. Signed informed consent

Exclusion criteria

1. Pre-existing acute kidney injury
2. Kidney transplantation
3. Off-pump heart surgery
4. Pregnancy
5. End stage renal disease
6. Pregnancy (female subjects of childbearing potential must have a negative serum pregnancy test)
7. Subjects with any kind of dependency on the investigator (e.g. any subject who is under direct supervision of the investigator/co-investigators or employed by the investigator/co-investigators) 8 Subjects held in an institution by legal or official order (e.g. subjects in jail, prison, juvenile offender facility, or treatment facility including those who are in hospitals, alcohol, and drug treatment facilities under court order, and individuals with psychiatric illnesses who have been committed involuntarily to an institution)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-03; Primary Completion 2017-02 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in serum metabolite profile of niacinamide | Baseline and days 1 through 4

SECONDARY OUTCOMES:
Changes from baseline in urine metabolite profile of niacinamide | Baseline and days 1 through 4

OTHER OUTCOMES:
Adverse events | From enrollment through day 4, and at day 30

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No